CLINICAL TRIAL: NCT04467905
Title: Multi-Centre, Placebo-Controlled, Phase 2 Study of Etripamil Nasal Spray (NS) for the Reduction of Ventricular Rate in Patients With Atrial Fibrillation.
Brief Title: ReVeRA-201: Etripamil in Atrial Fibrillation, Phase 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Milestone Pharmaceuticals Inc. (Other)
Collaborators: The Montreal Health Innovations Coordinating Center (MHICC) (Other); JSS Medical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSP-2017-5001
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; ventricular rate control; rapid ventricular rate; etripamil
MeSH Terms: conditions — Atrial Fibrillation | interventions — etripamil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Administration of placebo at the emergency department for an episode of atrial fibrillation
  Interventions: Drug: Placebo
- Etripamil (Experimental): Administration of 70 mg etripamil at the emergency department for an episode of atrial fibrillation
  Interventions: Drug: Etripamil

INTERVENTIONS:
Drug: Etripamil — The formulation of etripamil nasal spray consists of MSP-2017 (etripamil), water, acetic acid, disodium ethylene-diamine-tetra-acetic acid (EDTA), and sulfuric acid. The dose of etripamil to be evaluated in this study is 70 mg.
  Other Names: MSP-2017
  Arms: Etripamil
Drug: Placebo — The formulation of placebo nasal spray consists of water, sodium acetate, disodium, disodium ethylene-diamine-tetra-acetic acid (EDTA), and sulfuric acid to reproduce the same pH as the etripamil formulation.
  Arms: Placebo

SUMMARY:
Many patients with atrial fibrillation (AF) experience persistent tachycardia with episodes of rapid ventricular rate despite chronic treatment to reduce ventricular rate. The objectives of this study were to demonstrate the superiority of a nasal spray of etripamil over placebo in reducing ventricular rate in patients with AF; and to evaluate the safety and efficacy of etripamil nasal spray in participants with AF.

DETAILED DESCRIPTION:
This was a multi-center, randomized, double-blind, placebo-controlled study to evaluate the effects of etripamil nasal spray in participants with AF. This study included Screening, the Treatment Period (Screening and Treatment Period occur on the same day) and safety follow-up procedures.

Each participant received placebo or 70 mg of etripamil intranasally; treatment were randomized in a 1:1 ratio, to yield 50 evaluable participants with AF in 2 groups of 25.

Participants with AF were selected by the Investigator. The screening procedures included obtaining informed consent, a review of inclusion/exclusion criteria, a complete physical examination, and recording of any concomitant medications.

After screening procedures were complete, eligible participants were randomized to receive etripamil or placebo. Heart rate was measured continuously via Holter Electrocardiogram (ECG) from at least 10 minutes prior to dosing to 6 hours after study drug administration. Participants had to exhibit a rapid ventricular rate (≥110 bpm measured during 1 minute) on the Holter report prior to drug administration in order to receive the study drug. Beyond 60 minutes after study drug administration, medical care was offered in accordance with the standard of care and the participant was discharged from the clinic, while still wearing the Holter device.

Participants underwent a safety follow-up assessment and return the Holter device approximately 24 hours post-dose. Participants were contacted by phone 7 days post-dosing for safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

A participant was eligible for study participation if they met all of the following criteria:

1. Aged 18 years and over.
2. Provided written informed consent.
3. Participants with episodes of paroxysmal, persistent or permanent AF, presenting with AF and a ventricular rate ≥110 bpm, measured over 1 minute
4. Participants received appropriate antithrombotic therapy as per the applicable guidelines for atrial fibrillation management (e.g., Canadian Cardiovascular Society (CCS) guidelines / European Society of Cardiology (ESC) guidelines).

   1. Etripamil (a calcium channel blocker) was intended for acute rate control only. If rhythm control was desired (outside of the present protocol), anticoagulation as per guidelines could be started after the administration of study drug.

Exclusion Criteria:

A participant was excluded from the study if they met any of the following criteria:

1. Had evidence of atrial flutter (ECG) at presentation.
2. Had a history of stroke, transient ischemic attack (TIA) or peripheral embolism within the last 3 months.
3. Had received by IV route any of the following within one hour before study drug administration: flecainide, procainamide, digoxin, beta-blocker, or calcium channel blocker.
4. Had signs and symptoms of severe congestive heart failure at presentation (e.g. tachypnea, oxygen desaturation <90% unless due to known pulmonary disease, pulmonary rales, sign of peripheral hypoperfusion).
5. Hemodynamic instability, with systolic blood pressure <90 mmHg or diastolic blood pressure <60 mmHg.
6. Known uncorrected severe aortic or mitral stenosis.
7. Hypertrophic cardiomyopathy with outflow tract obstruction.
8. Had a history of second- or third-degree atrioventricular block.
9. Regular rhythm suggesting a complete atrioventricular block.
10. Had a history or evidence of torsades de pointes, sick sinus syndrome, or Brugada syndrome.
11. Evidence of acute coronary syndrome within the last 12 months except if participant was successfully revascularized.
12. Positive pregnancy test result at screening, and females of childbearing potential who did not agree to use adequate method of contraception for the duration of the study.
13. Had evidence of any clinically significant acute or chronic condition of the nasal cavity (e.g., rhinitis or deviated septum) which could have interfered with administration of the study drug in either or both nasal cavities.
14. Had a history of sensitivity to verapamil.
15. Had previously participated in a clinical study for etripamil.
16. Had a history of sensitivity to any components of the investigational product.
17. Had signs of alcohol or drug intoxication at the time of presentation which, in the opinion of the Investigator, would have impacted the validity of study results.
18. Was participating in another drug or device study, or had received an investigational drug or device within 30 days of Screening.
19. Had evidence of clinically significant cardiovascular, endocrine, gastrointestinal, hematologic, hepatic, immunologic, neurologic, oncologic, pulmonary, psychiatric, or renal disease or any other condition which, in the opinion of the Investigator, would have jeopardized the safety of the participant or impacted the validity of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Roy, M.D, Principal Investigator — Montreal Heart Institute (MHI)
Locations (18):
- Canada (11):
  - QEII HSC - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Hamilton Health Science, Hamilton, Ontario
  - PACE (Partners in Advanced Cardiac Evaluation), Newmarket, Ontario
  - Ottawa Hospital General & Civic Campus Research Institute, Ottawa, Ontario
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - CHU Montréal, Montreal, Quebec
  - CIUSSS du Nord-de-l'Île-de-Montréal - Hôpital du Sacré-Cœur, Montreal, Quebec
  - CISSS Bas-Saint-Laurent / Hôpital de Rimouski, Rimouski, Quebec
  - CISSS des Laurentides / Unité de recherche clinique, Saint-Jérôme, Quebec
  - CIUSSS de l'Estrie - CHU, Sherbrooke, Quebec
  - CISSS de Lanaudière - Hôpital Pierre-Le Gardeur, Terrebonne, Quebec
- Netherlands (7):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Jeroen Bosch Ziekenhuis Rijnstate Ziekenhuis, Arnhem
  - Slingeland Ziekenhuis, Doetinchem
  - Treant Zorggroep, Emmen
  - Elkerliek Ziekenhuis, Helmond
  - Franciscus Gasthuis, Rotterdam
  - Gelre Ziekenhuizen, Zutphen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camm AJ, Piccini JP, Alings M, Dorian P, Gosselin G, Guertin MC, Ip JE, Kowey PR, Mondesert B, Prins FJ, Roux JF, Stambler BS, van Eck J, Al Windy N, Thermil N, Shardonofsky S, Bharucha DB, Roy D. Multicenter, Phase 2, Randomized Controlled Study of the Efficacy and Safety of Etripamil Nasal Spray for the Acute Reduction of Rapid Ventricular Rate in Patients With Symptomatic Atrial Fibrillation (ReVeRA-201). Circ Arrhythm Electrophysiol. 2023 Dec;16(12):639-650. doi: 10.1161/CIRCEP.123.012567. Epub 2023 Nov 11. PMID 37950726

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with atrial fibrillation and ventricular rate =>110bpm over 1 minute were screened to participate in the study (first participant enrolled on 19-Nov-2020, last participant completed 10-Aug-2023). Overall, 87 participants were screened and from those, 69 participants were randomized. From those participants, 56 participants received etripamil or placebo.
Pre-assignment Details: Of the 69 participants randomized, 13 (18.8%) did not receive etripamil/placebo because of the following reasons: baseline heart rate <110bpm (n=5), converted to sinus rhythm (n=3), technical issue with Holter and ECGs were missing (n=3), hemodynamic instability (n=1), site misinterpretation of protocol (n=1).
Groups:
- Placebo: Participants randomized who received the placebo
- Etripamil: Participants randomized who received etripamil NS
- Randomized But Did Not Receive Drug: Participants randomized but did not receive placebo or etripamil
Period: Overall Study
Arm/Group | Placebo | Etripamil | Randomized But Did Not Receive Drug
Started | 29 | 27 | 13
Medication Was Administered | 29 | 27 | 0
Medication Was Not Administered | 0 | 0 | 13
Safety Population | 29 | 27 | 0
mITT Population | 29 | 27 | 0
Efficacy Population | 25 | 24 | 0
Completed | 29 | 27 | 0
Not Completed | 0 | 0 | 13
Not completed — Baseline heart rate <110 bpm | 0 | 0 | 5
Not completed — Conversion to SR | 0 | 0 | 3
Not completed — Technical issue with Holter ECG | 0 | 0 | 3
Not completed — Hemodynamic instability | 0 | 0 | 1
Not completed — Site misinterpretation of protocol | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety/mITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Etripamil | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Customized [Mean (Standard Deviation); unit: years] — Age at Informed Consent
  years
    Age at Informed Consent | 64.6 (10.5) | 64.6 (10.6) | 64.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 18 | 16 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 26 | 55
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 29 | 24 | 53
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Participant symptomatic during AF episode [Count of Participants; unit: Participants]
  No | 8 | 5 | 13
  Yes | 21 | 22 | 43
Type of AF [Count of Participants; unit: Participants] — Paroxysmal AF: AF that is intermittent and terminates within ≤7 days of onset. Persistent AF: AF that is continuous and sustains for >7 day and requires intervention.
  Permanent AF: AF that patient and clinician decide to stop further attempts to restore/maintain sinus rhythm.
  Participants
    Paroxysmal | 22 | 20 | 42
    Persistent | 5 | 5 | 10
    Permanent | 2 | 2 | 4
Participant had pacemaker [Count of Participants; unit: Participants]
  No | 28 | 27 | 55
  Yes | 1 | 0 | 1
AF diagnosis confirmed by ECG [Count of Participants; unit: Participants]
  No | 0 | 0 | 0
  Yes | 29 | 27 | 56
Systolic blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 125.6 (17.3) | 130.0 (19.8) | 127.7 (18.5)
Diastolic blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 85 (15.5) | 85.6 (18.6) | 85.3 (16.9)
Heart rate (bpm) [Mean (Standard Deviation); unit: bpm] | 134.9 (22.9) | 129.2 (13.0) | 132.1 (18.8)

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Reduction in Ventricular Rate, Measured on Holter Monitoring, Within 60 Minutes From Drug Administration.
Description: Baseline ventricular rate is defined as the average heart rate over 5 minutes immediately prior to drug administration.
  Nadir is defined as the lowest moving average heart rate over 5 minutes recorded in the 60 minutes post drug administration.
Time Frame: 60 minutes post drug administration
Population: The primary efficacy analysis was performed on the 49 participants in the Efficacy Population.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | Etripamil
Number analyzed (Participants) | 25 | 24
bpm
  Baseline Ventricular Rate (bpm) | 135.5 (13.9) | 130.3 (15.3)
  Nadir (bpm) | 130.7 (16.4) | 95.2 (23.7)
Statistical Analysis 1: Comparison: Placebo vs Etripamil; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -29.9, 95% CI 2-sided [-40.3 to -19.3] — The mean difference is the difference in adjusted means for the change between baseline value and nadir in the placebo group and the change between baseline and nadir in the etripamil group

ADVERSE EVENTS:
Time Frame: 7 days. Adverse events were monitored from Screening until study participation was complete after the final Follow-Up.
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product that did not necessarily have a causal relationship with the product.
  Untreated participants were not included in safety or efficacy analyses (were not included in safety or efficacy populations).
Arm/Group | Placebo | Etripamil
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/27
Serious Adverse Events (participants affected / at risk) | 4/29 | 1/27
Other Adverse Events (participants affected / at risk) | 18/29 | 23/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | Etripamil (N=27)
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | Etripamil (N=27)
Intracardiac thrombus (Cardiac disorders) | 2 | 0
Lacrimation increased (Eye disorders) | 5 | 8
Nasopharyngitis (Infections and infestations) | 0 | 2
Dizziness (Nervous system disorders) | 3 | 5
Headache (Nervous system disorders) | 0 | 3
Paraesthesia (Nervous system disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 11 | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 9
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Hot flush (Vascular disorders) | 1 | 2
Bradyarrhythmia (Cardiac disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT04467905/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT04467905/SAP_001.pdf